CLINICAL TRIAL: NCT01034228
Title: Exploratory Study to Evaluate the Effect of L-isoleucine Supplemented Oral Rehydration Solution in the Treatment of Acute Diarrhoea in Children and in Inducing Innate Immunity
Brief Title: Isoleucine Added ORS in Children With Diarrhoea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Georgetown University (Other); University Hospital, Basel, Switzerland (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-018
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2006-04

CONDITIONS: Acute Infectious Diarrhoea in Children
Keywords: Diarrhoea; L-isoleucine; children; ORS; Antibacterial peptide
MeSH Terms: conditions — Diarrhea | interventions — ORALIT; Isoleucine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoleucine (Active Comparator): Glucose ORS with L-Isoleucine
  Interventions: Other: ORS + Isoleucine
- ORS without Isoleucine (Placebo Comparator): ORS without Isoleucine for the treatment of diarrhoea in children
  Interventions: Other: ORS without Isoleucine

INTERVENTIONS:
Other: ORS + Isoleucine — ORS with Isolelucine for treatment of diarrhoeal in children
  Arms: Isoleucine
Other: ORS without Isoleucine — ORS without Isoleucine for the treatment of diarrhoea in children
  Arms: ORS without Isoleucine

SUMMARY:
Efforts are continuing to improve the efficacy of oral rehydration solution in terms of reducing the severity (stool volume) and duration of diarrhoea (enhancement of recovery). Antimicrobial peptides, produced by the epithelial cells, represent an important component of the innate immunity of all epithelial surfaces of the body including intestine. Induction of expression of antimicrobial peptides on epithelial cell surface, may thus hasten recovery from infectious diarrhoea. Isoleucine is an essential amino acid that is easily available and not very expensive, and its addition to oral rehydration solution might help early clearance of diarrhoeal pathogen by inducing secretion of antimicrobial peptide by the small intestinal epithelial cells. Additionally, it is expected to hasten recovery from diarrhoea by reestablishing the commensal bacteria. The aim of this pilot study is to assess if addition of isoleucine to oral rehydration solution induces secretion of antimicrobial peptide, help establish normal bacterial populations in the intestine, and favourably impacts the severity and duration of diarrhoea in young children. If the results are found encouraging, a therapeutic trial with adequate sample size would be justified.

DETAILED DESCRIPTION:
Globally, diarrhoea still accounts for 1.6 to 2.5 million deaths annually, and children in the developing world experience an average of 3 episodes of diarrhoea each year. Despite the decline in diarrhoeal mortality, it remains a leading cause of childhood morbidity and deaths [1]. Prevention of dehydration using appropriate home-made fluids or ORS solution, and correction of dehydration using ORS solution or intravenous fluid as indicated followed by maintenance of hydration using ORS solution, along with continuation of usual food including breastfeeding are most important elements of management of acute diarrhea. Antimicrobial therapy is recommended in the management of a few specific etiologic diarrhoeas such as severe cholera, shigellosis, invasive intestinal amoebiasis, and symptomatic giardiasis. The cost of therapy and more importantly the emergence of resistance pathogens are the major concerns for antimicrobial therapy for diarrhoea as for other bacterial infections.

ORS plays a major role in the treatment diarrhoeal diseases; however, it does neither reduce the severity nor the duration of diarrhoea, its major limitations. Efforts are continuing to overcome these limitations by developing newer formulations and delivery mechanisms e.g.

1. Changing/replacing the substrates (e.g. addition of alanine or glycine to glucose or replacing glucose by multodextrin and rice powder)
2. Reducing the concentration of glucose and sodium and thus osmolarity of ORS solution.

Alanine/glycine and rice powder containing ORS demonstrated some reduction in the stool output [2-5]. However, none of the formulations developed and tested till date demonstrated any beneficial effect on the duration of diarrhoea. Similarly, reduced osmolarity ORS has some beneficial effect on reducing the stool output and vomiting, and reducing failure of ORT mainly in children with non-cholera diarrhea, but did not have any effect on the diarrhoea duration [6]. The World Health Organization (WHO) and the United Nations Children Fund (UNICEF) have recently recommended routine use of the reduced-osmolarity ORS in the management of diarrhoeal diseases [7]; however, there are scopes to further improve its efficacy.

Antimicrobial peptides and innate immunity

Antimicrobial peptides represent an important component of the innate immune defenses of organisms ranging from plants to insects to humans. They are broad-spectrum, surface-active agents that kill microbes by forming pores in their membranes. Most have broad spectrum of activities against bacteria, viruses and fungi. In mammals, two major classes of antimicrobial peptides have been described- defensins and cathelicidins (LL-37). The defensins are a subclass of antimicrobial peptides, and in mammals, they are present in neutrophil granules where they are necessary for the non-oxidative killing of phagocytised microbes [8]. It is now well established that defensins are also produced at virtually all epithelial surfaces of mammals, including those of the skin, airways, gut, and urogenital tracts [9, 10]. Expression of some epithelial defensins is constitutive and contributes to a non-inflammatory antimicrobial barrier at the epithelial surface. Other defensins are inducible and highly expressed at sites of inflammation or infection [9, 11, 12]. Impairment of defensin functions increases susceptibility to infection of the airway in cystic fibrosis [13] and to enhanced Salmonella infection in the mouse intestinal tract [14]. In addition to their direct antimicrobial activities, Beta-defensins are chemotactic for memory T cells and dendritic cells, suggesting that they play an important role in the integration of the innate and acquired immune responses [15].

The molecular mechanisms underlying induction of epithelial defensins remain largely unexplored. Pattern-recognition receptors [16] likely play a critical role in this process, as has been shown in CD-14-mediated induction of Beta-defensins by bacterial lipopolysaccharide [17]. Whole heat-killed bacteria and fungi induce human Beta-defensins-2 in human keratinocytes, but the molecular basis of this response is not understood [11]. Inflammatory cytokines such as tumor necrosis factor Alpha (TNF) and IL-10 also induces Beta-defensins [18, 19]. Because pharmacological induction of defensins at epithelial barriers may have therapeutic utility, a search for novel molecules that could induce production of epithelial defensin, assessed by using cell-based assays, have long been underway. It has recently been observed that L-isoleucine and its analogues are highly specific Beta-defensin inducers in epithelial cells [20]. It has also been observed that when isoleucine is administered to animals (chicken), the gut flora shifts to the probiotic species, it stimulates paneth cells to secrete antimicrobial peptides in human intestinal tissue, and it causes a shift in gut flora leading to an increased numbers of Lactobacilli. (Manuscript, Ashida T & M Zasloff et al) in treatment of patients with Crohn's disease.

The above observations suggest a potential role of L-isoleucine in the management of infections of mucosal tissues including those in the gastrointestinal tract.

Antimicrobial peptides in Shigella infections

In 2001, researchers from ICDDRB and Karolinska Institute (BA) reported in Nature Medicine a down regulation of LL-37 and human Beta-defensin-1 (HBD-1) in the epithelial cells in diarrhoea caused by Shigella dysenteriae type I and other enteric bacteria [21]. This down regulation could be reproduced in vitro by using the cell lines U937 of monocyte origin and HT-29 of colonic epithelial origin, when infected with Shigella or plasmid DNA derived from Shigella. The down regulation can be an important immune escape mechanism for pathogens to avoid potent mucosal effector molecules such as antimicrobial peptides. Since antimicrobial factors drench the mucosal surfaces, it is conceivable that pathogenic bacteria down-regulate the front line defenses of humans as a part of their invasive process. Therefore, a novel approach will be to block this down-regulation or to take a therapeutic approach to up-regulate the production of endogenous antimicrobials. Recent studies have shown that short chain fatty acids (SCFA) can up-regulate expression of LL-37 in colonic epithelial cells, and among them sodium butyrate was the best inducer [22, 23]. Moreover, butyrate induces colonic cell differentiation that has been reported to be a key determinant of LL-37 expression in human colon epithelium [22]. However, it was shown that pathways other than those involved in cell differentiation are involved in the up-regulation of LL-37 with butyrate [23]. Butyrate is produced in the colon by fermentation of dietary fibre. Thus, there is a link between the normal gut flora and the expression of endogenous antibiotics. Additionally, SCFAs including butyrate has been shown to reduce clinical symptoms, and alter microbiological and pathological features in experimental Shigella infections in rabbit models [24]. Thus, a relationship between the severity of Shigella infections and mucosal levels of antimicrobial peptides is conceivable. Oral administration of sodium butyrate to rabbits infected with Shigella showed up-regulation of CAP-18 (rabbit homologue of LL-37) in the colonic epithelial cells with a concomitant reduction in shigella load in stool and clinical recovery (Raqib et al, manuscript accepted). Preventing down-regulation or enhancing antimicrobial peptide expression could provide an alternative treatment in protecting humans and animal livestock against bacterial pathogens. These studies may provide a basis for therapeutic manipulation of endogenous antimicrobial peptides including LL-37 expression in vivo using dietary substances or butyrate to strengthen the epithelial defense barrier. Therefore, we have initiated a clinical study in ICDDRB to evaluate the efficacy of butyrate enema in the treatment of shigellosis.

Butyrate has been shown to induce antimicrobial peptides in the colon; however; it can't be administered orally as such. Moreover, most of the acute diarrhoeal diseases are caused by infection of the small intestine. Isoleucine, an essential amino acid, might be a reasonable alternative for enhancing secretion of antimicrobial peptides from the paneth cells and other defense molecules from the upper small intestine (Manuscript, Ashida T & M Zasloff et al). This may help clear the pathogens, shift gut flora to a more "normal" commensal species distribution, and enhance recovery from infectious diarrhoea. Therefore, we hypothesize that use of L-isoleucine supplemented ORS solution will induce antimicrobial peptides and enhance clinical recovery of children with acute watery diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 months-36 months
2. Sex: only males, for precise separation of stool and urine
3. History of diarrhoea duration of <48 hours
4. Dehydration: some

Exclusion Criteria:

1. Diarrhoea due to Vibrio cholerae that requires antimicrobial therapy by dark field microscopy
2. Dysentery (blood in stool), which requires antimicrobial therapy
3. Concomitant infection(s) e.g. ARI, meningitis, and sepsis
4. History of taking antibiotics for the current diarrhoea episode
5. Severely malnourished children (Wt for length < 70%) or patients with edema

Ages: 6 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
1. Weight of abnormal (watery/liquid) stool for each 6-hour and 24-hour (day) of the study as well as cumulative weight until resolution of diarrhoea (maximum of 5 days) | 12 months

SECONDARY OUTCOMES:
1. ORS intake in different time periods, for each 6-hour and 24-hour (day) of the study as well as cumulative weight until resolution of diarrhoea (maximum of 5 days) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Hospital, ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Alam NH, Raqib R, Ashraf H, Qadri F, Ahmed S, Zasloff M, Agerberth B, Salam MA, Gyr N, Meier R. L-isoleucine-supplemented oral rehydration solution in the treatment of acute diarrhoea in children: a randomized controlled trial. J Health Popul Nutr. 2011 Jun;29(3):183-90. doi: 10.3329/jhpn.v29i3.7864. PMID 21766553